CLINICAL TRIAL: NCT00144365
Title: Comparison of Facility and Home-based ART Delivery Systems in Uganda
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: British Medical Research Council (Other Government); The AIDS Support Organization (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: CDC-NCHSTP-4371; 1U01PS000065-01 (NIH)
Record Dates: First submitted 2005-09-02; First posted 2005-09-05 (Estimated); Last update posted 2012-09-11 (Estimated); Status verified 2012-09

CONDITIONS: AIDS
Keywords: HIV; Africa; Adherence; HIV viral load; Sexual behavior; Voluntary counseling and testing
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Sexual Behavior | interventions — Antiretroviral Therapy, Highly Active

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Antiretroviral therapy

SUMMARY:
The study is a 3-year, randomized trial to compare ART delivery through two different models: a) ART delivered through health facilities by clinically qualified staff and b) home-based care in which lay workers, i.e. non-medically qualified people, play a major role in the ART delivery and clients are followed up at health facilities less frequently. The primary objective is to measure the effects of these strategies on HIV viral load. We will also examine the effects on treatment failure, disease progression, survival, adherence, family member HIV testing, sexual behavior, and cost-effectiveness.

DETAILED DESCRIPTION:
The study is a randomized trial to compare ART delivery through two different models: a) ART delivered through health facilities by clinically qualified staff and b) home-based care in which lay workers, i.e. non-medically qualified people, play a major role in the ART delivery and clients are followed up at health facilities less frequently. The primary objective is to measure the effects of these strategies on plasma HIV viral load. We will also examine the effects on treatment failure, disease progression, survival, adherence, family member HIV testing, sexual behavior, and cost-effectiveness.

The trial is conducted with The AIDS Support Organization (TASO) clinic in Jinja, Uganda. Randomization is conducted through geographic clusters, defined using sub-counties in the district, and stratified by distance from fixed health facilities, and urban/rural. Just over 800 participants, living in 40 clusters, will be recruited over a period of 3-6 months and followed-up over a period of 3 years.

ELIGIBILITY:
Inclusion Criteria:

HIV infection Plan to remain resident in the area for at least 12 months CD4 cell count <200 cells/mm3 or severe symptomatic HIV (WHO stage 3 or 4) Identify a medicine companion who will assist in adherence to ART treatment Age 18 years or above.

Exclusion Criteria:

Abnormal liver and renal function test results (AST or ALT ≥ 5x upper limit of normal Calculated creatinine clearance < 25 ml/min). The tests are conducted only in individuals in whom they are clinically indicated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1453 (Actual)
Dates: Start 2005-02; Primary Completion 2008-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
HIV viral load

SECONDARY OUTCOMES:
Medication adherence
Treatment failure
Morbidity
Survival
Sexual behavior
Family member HIV testing
cost-effectiveness

CONTACTS AND LOCATIONS:
Overall Officials: Heiner Grosskurth, MD, PhD, Principal Investigator — British Medical Research Council; Rebecca Bunnell, ScD, MEd, Principal Investigator — Centers for Disease Control and Prevention; Shabbar Jaffar, PhD, Principal Investigator — London School of Tropical Medicine and Hygeine; Alex Coutinho, MBChB, MSc, Principal Investigator — The AIDS Support Organization
Locations (1):
- The AIDS Support Organization, Jinja, Jinja, Uganda